CLINICAL TRIAL: NCT06617143
Title: Effects of Short-Term Conscious Awareness-Based Cognitıve Therapy Applied to Asthma Patients on Anxiety, Depression and Dyspnea
Brief Title: Effect of MBCT Applied to Asthma Patients on Anxiety, Depressıon and Dyspnea
Acronym: MBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ArdahanU-Şimsekli-DS-03
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Asthma; Mindfulness
Keywords: asthma; mindfulness-based cognitive therapy; anxiety; depression; dyspnea
MeSH Terms: conditions — Asthma; Anxiety Disorders; Depression; Dyspnea | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: pre-test post-test quasi-experimental design
Who Masked: Outcomes Assessor
Masking Description: Participants and researchers could not be blinded due to the natural course of the study and only the statistician was blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In this study, it is planned to apply MBCT to asthmatic inpatients in the patient room in groups of 2 or 3. This application is planned to continue for one hour.
  Interventions: Other: mindfulness-based cognitive therapy
- Control group (Active Comparator): No application will be made to the patients in the control group.
  Interventions: Other: routine treatment and care

INTERVENTIONS:
Other: mindfulness-based cognitive therapy — In this study, it is planned to apply MBCT to asthmatic inpatients in the patient room in groups of 2 or 3. This application is planned to continue for one hour.
  Arms: Experimental group
Other: routine treatment and care — routine treatment and care
  Arms: Control group

SUMMARY:
In this study, short-term MBCT will be applied to asthmatic patients receiving hospital treatment and its effects on anxiety, depression and dyspnea will be determined. A quasi-experimental study was planned for this purpose.

DETAILED DESCRIPTION:
In the study, cognitive behavioral therapy will be applied to the intervention group, which is determined as the experimental group, and a group of asthma patients who did not receive any application during the same periods will be included and the dyspnea, anxiety and depression levels of the patients in these two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years old, Inpatient treatment in the chest ward volunteer participants with no communication problems

Exclusion Criteria:

Under 18 years old, with communication problems, not willing to participate hospitalized with diseases other than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | Average of 1 week after completion of the intervention
  It will be evaluated with the Hospital Anxiety and Depression Scale.
Depression | Average of 1 week after completion of the intervention
  It will be evaluated with the Hospital Anxiety and Depression Scale.
Dyspnea | Average of 1 week after completion of the intervention
  It will be assessed with the Modified Medical Research Council (mMRC) Dyspnoea Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Derya ŞİMŞEKLİ, PhD, Principal Investigator — Ardahan University
Locations (1):
- Ardahan University, Ardahan, Ardahan, Turkey (Türkiye)

REFERENCES:
- [Background] FLETCHER CM. The clinical diagnosis of pulmonary emphysema; an experimental study. Proc R Soc Med. 1952 Sep;45(9):577-84. No abstract available. PMID 13003946
- [Background] Mahler DA, Weinberg DH, Wells CK, Feinstein AR. The measurement of dyspnea. Contents, interobserver agreement, and physiologic correlates of two new clinical indexes. Chest. 1984 Jun;85(6):751-8. doi: 10.1378/chest.85.6.751. PMID 6723384
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820